CLINICAL TRIAL: NCT02854748
Title: A Randomized, Open-label, Multiple Dosing, Crossover Study to Evaluate the Drug-drugs Interaction Between Lobeglitazone and Empagliflozin in Healthy Male Volunteers
Brief Title: Evaluate the Drug-drugs Interaction Between Lobeglitazone and Empagliflozin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19DDI16005
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; lobeglitazone

ARMS (6):
- Empagliflozin / Lobeglitazone / Empa.+Lobe. (Experimental): Period 1: Empagliflozin 25 mg QD for 5 days Period 2: Lobeglitazone 0.5 mg QD for 5 days Period 3: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg
- Empagliflozin / Empa.+Lobe. / Lobeglitazone (Experimental): Period 1: Empagliflozin 25 mg QD for 5 days Period 2: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days Period 3: Lobeglitazone 0.5 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg
- Lobeglitazone / Empagliflozin / Empa.+Lobe. (Experimental): Period 1: Lobeglitazone 0.5 mg QD for 5 days Period 2: Empagliflozin 25 mg QD for 5 days Period 3: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg
- Lobeglitazone / Empa.+Lobe. / Empagliflozin (Experimental): Period 1: Lobeglitazone 0.5 mg QD for 5 days Period 2: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days Period 3: Empagliflozin 25 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg
- Empa.+Lobe. / Empagliflozin / Lobeglitazone (Experimental): Period 1: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days Period 2: Empagliflozin 25 mg QD for 5 days Period 3: Lobeglitazone 0.5 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg
- Empa.+Lobe. / Lobeglitazone / Empagliflozin (Experimental): Period 1: Empagliflozin 25 mg + Lobeglitazone 0.5 mg QD for 5 days Period 2: Lobeglitazone 0.5 mg QD for 5 days Period 3: Empagliflozin 25 mg QD for 5 days
  Interventions: Drug: Empagliflozin 25mg; Drug: Lobeglitazone 0.5mg; Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg

INTERVENTIONS:
Drug: Empagliflozin 25mg — Empagliflozin 25 mg QD for 5 days
Drug: Lobeglitazone 0.5mg — Lobeglitazone 0.5mg QD for 5 days
Drug: Empagliflozin 25mg/Lobeglitazone 0.5mg — Empagliflozin 25 mg + Lobeglitazone 0.5mg QD for 5 days

SUMMARY:
This study is a randomized, open-label, multiple dosing, crossover study to evaluate the drug-drugs interaction between Lobeglitazone and Empagliflozin in healthy male volunteers

DETAILED DESCRIPTION:
To healthy male subjects of 30, following treatments are administered dosing in each 3 period(Lobeglitazone or Empagliflozin or Lobe.+Empa.) and wash-out period is a minimum of 7 days.

Test Drug 1: Lobeglitazone 0.5mg 1T

Test Drug 2: Empagliflozin 25mg 1T

Pharmacokinetic blood samples are collected up to 24hrs.

Safety, pharmacokinetic and the drug-drugs interaction are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy person whose age is in between 19 to 45 during the screening tests
2. Whose weight is more than 55 kg, BMI is over 18.5 and under 29.9 during the screening test. (BMI (kg/m2) = weight (kg) / {height (m)}2)
3. A male with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening tests
5. The participants must have an ability and willingness to participate throughout the entire trials

Exclusion Criteria:

1. A person who has a history of clinically significant cardiovascular, respiratory, liver, kidney, endocrine system, immune system, urinary system diseases, blood-tumor diseases, mental illness.
2. Who had a history of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy)
3. Who has a history of hypersensitivity reactions to Empagliflozin or Lobeglitazone or similar series or other excipient ingredients (aspirin, fibrate, antibiotics, etc.)
4. A person whose electrocardiogram value includes QTc > 450 msec, PR interval > 200 msec, QRS duration > 120 msec after screening, or who show clinically significant opinion.
5. Who falls under the following results

   1. Liver Function Test (AST, ALT) are exceeded over 1.5x the upper limit of the normal range
   2. eGFR < 60mL/min/1.73m2
6. Who shows the vital sign values of more than 150 mmHg or less than 90 mmHg in systolic pressure or more than 95 mmHg or less than 60 mmHg in diastolic blood pressure
7. Who has history of drug abuses or shows a positive result in the urinary drug screen
8. Who took any prescribed drugs, medicinal plants within the 2 weeks before the first day of dosing or takes any over-the-counter drugs or vitamin supplements within 1 week (but, if other conditions are met, they can still participate in the clinical test through the researcher's judgment)
9. Who took other investigational drugs or bioequivalence drugs within 3 months before the first day of dosing
10. Who participated in whole blood donation within 2 months before the first of dosing, or platelet donations within 1 months. Who received blood a month before the first day of dosing
11. Who constantly drinks alcohol (over 21 units/week, 1 unit = 10 g of pure alcohol) or cannot stop drinking alcohol during the clinical test.
12. Who smokes more than 10 cigarettes per day within 3 months , or who cannot quit smoking when hospitalized
13. Who cannot limit intake of grapefruit or grapefruit containing foods in 48hrs from the first dosing of clinical testing drug to collect pharmacokinetic blood samples
14. Who absorb caffeinated drinks (coffee, tea (black or green tea), soda, coffee flavored milk, energy drinks, etc.) or cannot stop absorbing them 24 hours before hospitalization until discharging
15. Not using a reliable contraception, planning a pregnancy during the study
16. Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders
17. Person who is not determined unsuitable to participate in this test by the researchers

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
AUC0-t,ss of Empagliflozin | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
Cmax,ss of Empagliflozin | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
AUC0-t,ss of Lobeglitazone | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
Cmax,ss of Lobeglitazone | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours

SECONDARY OUTCOMES:
Tmax,ss of Empagliflozin | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
t1/2,ss of Empagliflozin | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
AUCinf of Empagliflozin | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
Tmax,ss of Lobeglitazone | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
t1/2,ss of Lobeglitazone | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours
AUCinf of Lobeglitazone | Day 1, 2, 3, 4 (Day 12 - 15, Day 23 - 26): 0 hour, Day 5 (Day 16, Day 27): 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dong A University Hospital, Seo-gu, Busan, South Korea

REFERENCES:
- [Derived] Kim YK, Hwang JG, Park MK. No Relevant Pharmacokinetic Drug-Drug Interaction Between the Sodium-Glucose Co-Transporter-2 Inhibitor Empagliflozin and Lobeglitazone, a Peroxisome Proliferator-Activated Receptor-gamma Agonist, in Healthy Subjects. Drug Des Devel Ther. 2021 Apr 28;15:1725-1734. doi: 10.2147/DDDT.S302215. eCollection 2021. PMID 33953542